CLINICAL TRIAL: NCT05868213
Title: ERP Studies of Acute Influences of THC and CBD on Memory Encoding and Retrieval Processes: Experiment 1
Brief Title: Cannabis Observations on Brain Waves, Retrieval, and Attention: Experiment 1
Acronym: COBRA
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, L. Cinnamon Bidwell, Assistant Professor, University of Colorado, Boulder
Other Study IDs: 20-0309: Experiment 1; R01DA052431 (NIH)
Record Dates: First submitted 2023-04-11; First posted 2023-05-22 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cannabis; Memory; Electroencephalography
Keywords: Cannabis; Marijuana; Memory; Event-related potential; Electroencephalography; THC; CBD; Verbal learning; Episodic memory
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected for cannabinoid quantification and DNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cannabis (smoked flower) — Self-Directed Use (ad-libitum)

SUMMARY:
This study investigates the impact of ∆9-tetrahydrocannabinol (THC) and cannabidiol (CBD) on recognition memory in healthy, regular cannabis users. Participants complete the same recognition memory task after self-administering one of three different strains of cannabis flower one day and while not intoxicated another day. Event-related potentials (ERPs) are measured via electroencephalogram (EEG) during the recognition memory task. Blood is collected to quantify THC and CBD exposure. Participants also complete self-report measures of medical history, sleep quality, subjective cognitive function, physical activity, psychological functioning, substance use, and acute drug effects.

DETAILED DESCRIPTION:
Previous research has established cannabis's harmful cognitive impact, with particularly robust and consistent effects in the domain of verbal episodic memory. However, prior work has not sufficiently considered that the memory effects of cannabis are the compound action of different cannabinoids, which vary in their pharmacology and effects. Specifically, CBD, a non-psychotomimetic component of cannabis (doesn't produce a "high"), is thought to have cognitively protective properties and may mitigate some of the harmful effects of THC. Further, few prior studies have tested the effects of high potency strains that are commonly available.

This study tests the effects of commercially available cannabis flower strains on recognition memory performance and ERPs that are related to different underlying memory processes in healthy, regular cannabis users. An episodic memory task is used to assess recognition memory, which asks participants to discriminate between previously studied and non-studied items using words as stimuli. Participants complete the same memory task while intoxicated one day and not intoxicated another day. A THC-dominant, a CBD-dominant, and a strain containing both THC and CBD are included in the study. Participants self-administer one of the three cannabis strains prior to memory encoding and retrieval.

Blood is collected to determine THC and CBD exposure, as well as to explore how genetic variation in genes related to cannabinoid metabolism, cannabis-related behavior, and neurocognitive function associate with memory function before and after cannabis use. Participants also complete self-report measures of medical history, sleep quality, subjective cognitive function, physical activity, psychological functioning, substance use, and acute drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 21 and 40 and provide informed consent.
* Must be right-handed (Laterality Quotient > 60 on Edinburgh Handedness Inventory - Short Form).
* Must use cannabis at least 4 days during the month.
* Must be a cannabis user for at least a year.
* Must self-report not using other illicit recreational drugs (e.g., cocaine, benzodiazepines (non-prescription), opiates (non-prescription), MDMA, sedatives, or methamphetamine) in the past 30 days.
* Must not test positive on a urine toxicology test for drugs of abuse.
* Must not be using psychotropic medications, however anti-depressant, non-benzodiazepine anti-anxiety, and ADHD medications are ok. ADHD medication users must be willing to abstain from ADHD medication use on appointment days.
* Must not be a regular tobacco user (≤4 days per week; cigarette, E-cigs, or smokeless).
* Must not have used caffeine or tobacco (cigarette, E-cigs, or smokeless) for 4 hours prior to appointments.
* Must have a breath alcohol level of 0 to sign consent form.
* Must not be actively seeking or in treatment for any substance use disorder.
* Female subjects must not be or trying to become pregnant.
* Must not be in treatment for psychotic disorder or bipolar disorder; or have a history with these disorders.
* Must not have any physical characteristics (e.g., thick hair, head size exceeding the limit of the net, dyed hair) or experience any technical difficulties during testing that result in a poor-quality EEG recording.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Difference in ERP amplitude | intoxicated session and not-intoxicated session
  Electroencephalography is used to quantify FN400 and parietal ERP effects.
Difference in recognition memory performance | intoxicated session and not-intoxicated session (about 1 week)
  Accuracy and reaction time will be used to assess task performance.

SECONDARY OUTCOMES:
Difference in Flanker Task performance | intoxicated session and not-intoxicated session (about 1 week)
  Accuracy and reaction time will be used to assess task performance.
Difference in Flanker Task ERPs | intoxicated session and not-intoxicated session (about 1 week)
  Electroencephalography is used to quantify ERN effects.
Change in Positive and Negative Affect Schedule (PANAS) | before and after acute cannabis use (about 30 minutes)
  The PANAS is Self-report measurement of positive and negative affect.
Change in Drug Effects Questionnaire (DEQ) | before and after acute cannabis use (about 30 minutes)
  The DEQ is a visual analogue scale of measure of acute drug effects.
Change in Addiction Research Center Inventory (ARCI-M) | before and after acute cannabis use (about 30 minutes)
  The ARCI-M is a self-report measure of subjective effects of marijuana.
Change in Marijuana Craving Questionnaire | before and after acute cannabis use (about 30 minutes)
  The Marijuana Craving Questionnaire is a self-report measure of marijuana craving.
Change in Profile of Mood States (POMS) | before and after acute cannabis use (about 30 minutes)
  The POMS is a self-report measure of mood.
Change in Alcohol Craving Questionnaire | before and after acute cannabis use (about 30 minutes)
  The Alcohol Craving Questionnaire is a self-report measure of alcohol craving.
Change in State Adapted Paranoia Checklist-Brief (SAPC-B) | before and after acute cannabis use (about 30 minutes)
  The SAPC-B is a self-report measure of paranoia.
Difference in circulating cannabinoids | baseline, intoxicated session, and not-intoxicated session (about 3 weeks)
  Blood levels of THC and CBD will be quantified.

OTHER OUTCOMES:
Exploratory: Associations between genes related to cannabinoid metabolism, cannabis-related behavior, and neurocognitive function with ERPs and recognition memory performance | baseline, intoxicated session, and not-intoxicated session (about 3 weeks)
  DNA samples are collected from a baseline blood sample.
Exploratory: Moderation of primary effects by baseline health and psychological functioning | baseline, intoxicated session, and not-intoxicated session (about 3 weeks)
  Baseline health and psychological function include measures of sleep quality, affective symptoms, and substance use history.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Curran, PhD, Principal Investigator — University of Colorado, Boulder; L. Cinnamon Bidwell, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Center for Innovation and Creativity, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: More information — https://www.colorado.edu/center/cuchange/research